CLINICAL TRIAL: NCT03399032
Title: Pharmacokinetics of Caspofungin in Critically Ill Patients
Brief Title: Pharmacokinetics of Caspofungin
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Other Study IDs: KE-0254/330/2017
Record Dates: First submitted 2018-01-07; First posted 2018-01-16 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock; Fungal Infection; Critical Illness
Keywords: caspofungin; pharmacokinetics
MeSH Terms: conditions — Shock, Septic; Mycoses; Critical Illness | interventions — Caspofungin; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients' arterial blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caspofungin: Each patient will receive: caspofungin i.v. once daily ( 70 mg on the first day, 50 mg on the 2 and 3 day
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Each patient will receive: caspofungin i.v. once daily ( 70 mg on the first day, 50 mg on the 2 and 3 day
  Blood samples (3 mL) will be collected 2, 4, 8, 12 and 24 hours after each dose of caspofungin for 3 consecutive days.
  Other Names: blood collection

SUMMARY:
The objective of this study is to describe the pharmacokinetics of standard doses of caspofungin in critically ill patients.

DETAILED DESCRIPTION:
This is a prospective observational study performed on critically ill patients. Inclusion criteria are: severe sepsis on admission requiring broad-spectrum antibiotics. Both medical and surgical patients will be included. Any type of infections will be included (pulmonary, abdominal, urinary tract, etc.) Antibiotics regimen includes: broad spectrum anti-bacterial antibiotics plus caspofungin (70 mg i.v. on the first day day, and 50 mg i.v. on the consecutive days, once daily.

Blood samples (3 mL) will be collected 2, 4, 8,12 and 24 hours after each dose of caspofungin for 3 consecutive days. The standard arterial canula will be used to obtain samples.

30 minutes after each sample collection, blood will be centrifuged for 10 minutes at 3,000 rpms. Subsequently, supernatant will be collected and frozen.

Serum caspofungin concentration will be measured with high performance liquid chromatography.

Each patient's hemodynamics parameters will be recorded with the use of transpulmonary thermodilution technique (PICCO). Other therapies i.e.: ventilatory support, sedation, an antifungal agent will be given as required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require ICU treatment due to severe sepsis age
* 18-80 years
* an eligible consent obtained from the patient or his/her attendant

Exclusion Criteria:

* allergy to caspofungin
* lack of consent to participate in the study
* age of patients below 18 or above 80 years

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU due to severer sepsis recognition. Both medical and surgical patients will be included. Any site of infection will be treated in the manner.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Serum concentration of caspofungin | 72 hours for each patient from the tigecycline treatment initiation
  Samples obtain from ICU patients 2, 4, 8 12 and 24hours after each dose of caspofungin for 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- II Department of Anesthesia and Intensive Care, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borsuk-De Moor A, Sysiak-Slawecka J, Rypulak E, Borys M, Piwowarczyk P, Raszewski G, Onichimowski D, Czuczwar M, Wiczling P. Nonstationary Pharmacokinetics of Caspofungin in ICU Patients. Antimicrob Agents Chemother. 2020 Aug 20;64(9):e00345-20. doi: 10.1128/AAC.00345-20. Print 2020 Aug 20. PMID 32601169